CLINICAL TRIAL: NCT06127901
Title: Prevalence and Risk Factors for Postoperative Delirium 48 Hours After Surgery: Multicenter Cohort Study.
Brief Title: Prevalence and Risk Factors for Postoperative Delirium 48 Hours After Surgery
Acronym: DELPO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Other Study IDs: DELPO
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: Patients over 18 years of age undergoing urgent and scheduled surgery requiring hospital admission, under any type of anaesthesia.
  Interventions: Procedure: Any surgery under any type of anaesthesia.

INTERVENTIONS:
Procedure: Any surgery under any type of anaesthesia. — Any surgery under any type of anaesthesia.

SUMMARY:
To determine the overall prevalence of postoperative delirium (POI) and its association with different risk factors in order to establish prevention plans to reduce its incidence and/or duration in Spanish hospitals.

To this end, patients over 18 years of age who underwent urgent and scheduled surgery requiring hospital admission under any type of anaesthesia during two specific days will be recruited and pre-, intra- and postoperative data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age undergoing urgent and scheduled surgery requiring hospital admission, under any type of anaesthesia.

Exclusion Criteria:

* Presence of pre-surgical delirium.
* Outpatient surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age undergoing urgent and scheduled surgery requiring hospital admission, under any type of anaesthesia.
Sampling Method: Probability Sample
Enrollment: 1535 (Estimated)
Dates: Start 2023-11-14 (Estimated); Primary Completion 2024-01-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Postoperative Delirium in Spanish hospitals. | 2 days
  To determine the overall prevalence of Postoperative Delirium in Spanish hospitals.

SECONDARY OUTCOMES:
Prevalence of Postoperative Delirium by surgical speciality. | 2 days
  To determine the prevalence of Postoperative Delirium by surgical speciality.
Risk factors on the prevalence of Postoperative Delirium | 2 days
  Determine the influence of risk factors on the prevalence of Postoperative Delirium

CONTACTS AND LOCATIONS:
Locations (63):
- Spain (63):
  - Hospital Complex of Ferrol, Ferrol, A Coruña
  - Santiago de Compostela University Clinical Hospital, Santiago de Compostela, A Coruña
  - General University Hospital of Elche, Elche, Alicante
  - University Hospital of Son Espases, Palma de Mallorca, Balearic Islands
  - Germans Trials i Pujol Hospital, Badalona, Barcelona
  - University Hospital of Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Parc Taulí Hospital, Sabadell, Barcelona
  - Marqués de Valdecilla University Hospital, Santander, Cantabria
  - Comarcal Hospital of Castellón, Vinaròs, Castellón
  - General University Hospital of Castellón, Castellon, Castelló
  - Donostia University Hospital, Donostia / San Sebastian, Giguzkoa
  - Doctor Negrín University Hospital, Las Palmas de Gran Canaria, Las Palmas
  - Public Hospital of Mariña, Burela de Cabo, Lugo
  - Regional Hospital of Monforte de Lemos, Monforte de Lemos, Lugo
  - Príncipe de Asturias University Hospital, Alcalá de Henares, Madrid
  - Henares Hospital, Coslada, Madrid
  - Fuenlabrada University Hospital, Fuenlabrada, Madrid
  - Puerta de Hierro University Hospital, Majadahonda, Madrid
  - University Hospital of Móstoles, Móstoles, Madrid
  - Quirónsalud University Hospital, Pozuelo de Alarcón, Madrid
  - Infanta Sofía University Hospital, San Sebastián de los Reyes, Madrid
  - Quirónsalud Valle del Henares Hospital, Torrejón de Ardoz, Madrid
  - Cabueñes University Hospital, Gijón, Principality of Asturias
  - Central University Hospital of Asturias, Oviedo, Principality of Asturias
  - Canarias University Hospital, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Francesc de Borja Regional Hospital, Gandia, Valencia
  - Manises Hospital, Manises, Valencia
  - Cruces University Hospital, Barakaldo, Vizcaya
  - Basurto University Hospital, Bilbao, Vizcaya
  - Hospital Complex of A Coruña, A Coruña
  - San Juan University Hospital, Alicante
  - Sant Joan University Hospital of Alacant, Alicante
  - University Hospital of Badajoz, Badajoz
  - Santa Creu i Sant Pau Hospital, Barcelona
  - Clinic Hospital of Barcelona, Barcelona
  - University Hospital of Burgos, Burgos
  - San Pedro de Alcántara Hospital, Cáceres
  - Reina Sofía Hospital, Córdoba
  - Infanta Margarita Hospital, Córdoba
  - Josep Trueta University Hospital, Girona
  - San Cecilio University Hospital, Granada
  - Hospital of León, León
  - Lucus Augusti Universitary Hospital, Lugo
  - San José and Santa Adela Cruz Roja Central Hospital, Madrid
  - La Princesa University Hospital, Madrid
  - Infanta Leonor University Hospital, Madrid
  - San Carlos Clinical Hospital, Madrid
  - 12 Octubre University Hospital, Madrid
  - La Paz Universitary Hospital, Madrid
  - La Paz University Hospital, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Complex of Ourense, Ourense
  - Montecelo Hospital, Pontevedra
  - University Hospital of Salamanca, Salamanca
  - Virgen de la Macarena University Hospital, Seville
  - Clinic Hospital of Valencia, Valencia
  - General University Hospital of València, Valencia
  - Doctor Peset Universitary Hospital, Valencia
  - La Fe University and Polytechnic Hospital, Valencia
  - University Clinical Hospital of Valladolid, Valladolid
  - Ribera Povisa Hospital, Vigo
  - Álvaro Cunqueiro University Hospital, Vigo
  - Miguel Servet University Hospital, Zaragoza